CLINICAL TRIAL: NCT06090318
Title: A Phase 1b/2Study of Milademetan in Combination With Atezolizumab in Patients With Advanced Solid Tumors With CDKN2A Loss (MANTRA-4)
Brief Title: Milademetan in Combination With Atezolizumab in Patients With Advanced Solid Tumors With CDKN2A Loss
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Rain Oncology Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAIN-3204
Record Dates: First submitted 2022-11-14; First posted 2023-10-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Advanced Solid Tumor; CDKN2A; NSCLC; Urothelial Carcinoma Bladder; Melanoma; Pancreas Adenocarcinoma; HNSCC; Renal Cell Carcinoma; Mesothelioma; Gastric Cancer
Keywords: CDKN2A; WT TP53; Advanced Solid Tumor; Wild-type P53
MeSH Terms: conditions — Melanoma; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Renal Cell; Mesothelioma; Stomach Neoplasms | interventions — milademetan; atezolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Milademetan (RAIN-32) in Combination With Atezolizumab (Experimental): Milademetan (RAIN-32): 260 mg orally on 3 consecutive day sets with a minimum of 14 days and a maximum of 21 days between the first day of each 3- day dosing set.
  Atezolizumab: Atezolizumab IV infusion is to be administered on Day 1 of each 28- day cycle.
  Interventions: Drug: Milademetan; Drug: Atezolizumab

INTERVENTIONS:
Drug: Milademetan — 260 mg once daily orally on 3 consecutive day sets with a minimum of 14 days and a maximum of 21 days between the first day of each 3- day dosing set.
  Other Names: RAIN-32
Drug: Atezolizumab — 1680mg administered every 4 weeks
  Other Names: TECENTRIQ

SUMMARY:
This is an open-label, single-arm, Phase 1b/2 study designed to evaluate the safety, tolerability, and preliminary efficacy of milademetan in combination with atezolizumab in patients with advanced solid tumors with confirmed homozygous CDKN2A loss and WT TP53 who have progressed on or are refractory to prior PD-1/PD-L1 inhibitor therapy and who, in the opinion of the Investigator, are unlikely to tolerate or derive clinically meaningful benefit from other therapy.

This study will determine the recommended dose of milademetan when given in combination with atezolizumab (the combination RP2D) using a dose de-escalation safety assessment cohort (Phase 1b).

Following identification of the combination RP2D, the safety profile and preliminary anti-tumor activity of the combination RP2D will be evaluated in a larger population in a dose expansion cohort (Phase 2).

DETAILED DESCRIPTION:
Up to 30 patients will be enrolled, 3 to 18 patients in the safety assessment cohort and 12 to 27 patients in the dose expansion cohort.

ELIGIBILITY:
Key Inclusion Criteria:

* Has a histologically confirmed, advanced solid tumor that has progressed on prior therapy with an anti-PD-1/L1 inhibitor administered as either monotherapy or in combination with other therapies
* Has documented homozygous CDKN2A loss and Wild-Type TP53
* Confirmation of available tumor tissue collected within 5 years of enrollment
* Measurable tumor lesions per RECIST 1.1
* Estimate life expectancy of at least 6 months
* ECOG PS of 0 or 1
* Resolution of clinically relevant toxic effect of prior anti-cancer therapies Note: AEs from prior therapy must resolve to Grade ≤ 1 per the NCI CTCAE version 5.0, except for peripheral neuropathy, which must resolve to Grade ≤ 2, and alopecia
* Adequate bone marrow, renal and hepatic function

Key Exclusion Criteria:

* Has received prior treatment with any MDM2 inhibitor; prior treatment with atezolizumab is allowed except if the patient discontinued due to toxicity
* Has a history of any Grade 3 or 4 immune-related toxicities to a prior checkpoint inhibitor treatment or history of treatment discontinuation with prior checkpoint inhibitor use due to toxicity

  * Endocrinopathies which are stable with appropriate hormonal supplementation consistent with other eligibility parameters
  * Dermatologic events which have resolved to Grade ≤ 1 on stable medication, as appropriate, and consistent with other eligibility parameters
* Treatment with systemic immunosuppressive medication, including but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and antitumor necrosis factor agents, within 2 weeks prior to the first dose of study treatment or anticipation of need for systemic immunosuppressive medication during the course of the study
* Has an uncontrolled infection within the 7 days prior to Screening
* Has undergone treatment with therapeutic oral or IV antibiotics within 2 weeks prior to first dose of study treatment
* Has known active central nervous metastases and/or carcinomatous meningitis. Note: Patients who require steroids for brain metastases must be on a stable or tapering dose of corticosteroids for at least 2 weeks before the first dose of study treatment. If applicable, patients must complete stereotactic radiosurgery 7 days before, and spinal or whole brain radiotherapy 21 days before, their first dose of study treatment
* Has as other primary malignancies that have required systemic antineoplastic treatment within 2 years prior to Screening, except for localized cancers that have apparently been cured (eg, nonmelanoma skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast) and will not interfere with the study outcomes
* Has uncontrolled or significant cardiovascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-05-19 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
The number of participants with treatment related AEs meeting DLT-defined criteria assessed by CTCAE v5.0 when receiving milademetan in combination with atezolizumab in patients with advanced solid tumors with HZ CDKN2A loss and WT TP53 | 4 months
The appropriate dose of milademetan in combination with atezolizumab based on the number of participants with DLT-defined adverse events assessed by CTCAE v5.0 criteria | 4 months
Treatment emergent AE of the identified RP2D of milademetan in combination with atezolizumab in patients with advanced solid tumors with HZ CDKN2A loss and WT TP53 | 24 months

SECONDARY OUTCOMES:
Objective response rate (ORR) | 24 months
  ORR, defined as the percentage of patients who achieve a confirmed CR or PR
Duration of response (DOR) | 24 months
  DOR, defined as the time from the date of first response (CR or PR) to the date of radiologically demonstrated disease progression, or death due to any cause
Disease control rate (DCR) | 24 months
  DCR, defined as the percentage of patients who achieve CR, PR, or SD for ≥ 16 weeks
Progression Free Survival (PFS) | 24 months
  PFS, defined as the time from the date of first dose to the earliest date of the first objective documentation of radiographic disease progression, or death due to any cause
Growth Modulation Index (GMI) | 24 months
  GMI: The GMI will be determined using the ratio of time to progression (TTP) with nth line of therapy (TTPn; here defined milademetan plus atezolizumab) to the most recent prior line of therapy (TTPn-1)
Pharmacokinetics Cmax | Initiation of study treatment through milademetan dose 13, an average of 3 months
  PK: maximum plasma concentration (Cmax) of milademetan
Pharmacokinetics AUC | Initiation of study treatment through milademetan dose 13, an average of 3 months
  PK: area under the plasma concentration-time curve (AUC)
Pharmacokinetics Tmax | Initiation of study treatment through milademetan dose 13, an average of 3 months
  PK: Time to reach maximum plasma concentration of milademetan